CLINICAL TRIAL: NCT03808610
Title: Phase I/II Study of the Combination of Low-Intensity Chemotherapy and Venetoclax (ABT-199) in Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia (ALL)
Brief Title: Low-Intensity Chemotherapy and Venetoclax in Treating Patients With Relapsed or Refractory B- or T-Cell Acute Lymphoblastic Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0629; NCI-2018-03360 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0629 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-01-16; First posted 2019-01-17 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Recurrent B Acute Lymphoblastic Leukemia; Recurrent T Acute Lymphoblastic Leukemia; Refractory B Acute Lymphoblastic Leukemia; Refractory T Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Methotrexate; merphos; nelarabine; pegaspargase; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; venetoclax; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (venetoclax, vincristine, cyclophosphamide) (Experimental): See Detailed Description.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Methotrexate; Drug: Nelarabine; Drug: Pegaspargase; Drug: Prednisone; Biological: Rituximab; Drug: Venetoclax; Drug: Vincristine

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Nelarabine — Given IV
  Other Names: 2-Amino-6-methoxypurine arabinoside; 506U78; Arranon; Compound 506U78; GW506U78
Drug: Pegaspargase — Given IV
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
Drug: Vincristine — Given IV
  Other Names: LEUROCRISTINE; VCR; Vincrystine

SUMMARY:
This phase I/II trial studies the side effects and best dose of venetoclax and how well it works in combination with low-intensity chemotherapy in patients with B- or T-cell acute lymphoblastic leukemia that has not responded to treatment or that has come back. Venetoclax may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, including vincristine, cyclophosphamide, dexamethasone, rituximab, methotrexate, and cytarabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving venetoclax with low-intensity chemotherapy may work better in treating patient with B- or T-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) and dose-limited toxicities (DLTs) of venetoclax in combination with low-intensity chemotherapy in patients with relapsed/refractory acute lymphoblastic leukemia (ALL) (Phase I).

II. Evaluate the overall response rate (complete response [CR] + CR with inadequate count recovery [CRi]) of the regimen after 2 cycles. (Phase II)

SECONDARY OBJECTIVES:

I. Evaluate other clinical efficacy endpoints (minimal residual disease [MRD] negativity, duration of response [DOR], event-free survival [EFS] and overall survival [OS]).

II. Determine the safety of the combination regimen.

EXPLORATORY OBJECTIVES:

I. To correlate apoptotic protein expression and Bcl-2 dependency on response and resistance to the combination regimen.

OUTLINE: This is a phase I, dose-escalation study of venetoclax, followed by a phase II study.

CHEMOTHERAPY AND VENETOCLAX:

CYCLE 1: Patients receive venetoclax orally (PO) once daily (QD) on days 1-21, vincristine intravenously (IV) over 15 minutes on days 7 and 17, cyclophosphamide IV twice daily (BID) over 3 hours on days 7-9, and dexamethasone IV over 30 minutes or PO QD on days 7-10 and 17-20. Patients may also receive rituximab IV over 4-6 hours on days 7 and 17 per physician discretion.

CYCLES 2, 4, 6, and 8: Patients receive venetoclax PO QD on days 1-21, methotrexate IV over 24 hours on day 1, and cytarabine IV BID over 3 hours on days 2 and 3. Patients may also receive rituximab IV over 4-6 hours on days 1 and 8 per physician discretion.

CYCLES 3, 5, and 7: Patients receive venetoclax PO QD on days 1-21, cyclophosphamide IV BID over 3 hours on days 1-3, vincristine IV over 15 minutes on days 1 and 11, and dexamethasone IV over 30 minutes or PO QD on days 1-4 and 11-14. Patients may also receive rituximab IV over 4-6 hours on days 1 and 11 per physician discretion.

T-CELL ALL: After the first 4 cycles, patients receive nelarabine IV over 2 hours on days 1-5 and pegaspargase IV over 2 hours on day 5. Cycles repeat every 28 days for 2 cycles (after cycle 4 and 5) in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients may receive prednisone PO QD on days 1-5, vincristine IV over 15 minutes on day 1, and venetoclax, PO QD on days 1-21. Cycles repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

T-CELL ALL (MAINTENANCE THERAPY): After the first 5 cycles of maintenance therapy, patients who received nelarabine and pegaspargase will receive nelarabine IV QD over 2 hours on days 1-5 and pegaspargase IV over 2 hours on day 5 during maintenance cycles 6 and 7 instead of prednisone, vincristine, and venetoclax.

After completion of study treatment, patients are followed up for 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of one of the following

   1. Patients ≥ 18 years of age with relapsed/refractory B- or T-cell ALL (for phase II only)
   2. Patients ≥ 60 years of age with previously untreated B- or T-cell ALL. Patients <60 years of age may be enrolled if they are considered unfit for intensive chemotherapy
   3. Patients ≥ 60 years of age with previously treated B- or T-cell ALL who received 1-2 courses of any frontline chemotherapy. Patients <60 years of age may be enrolled if they are considered unfit for intensive chemotherapy

      * If they achieved CR/CRi, they are assessable only for event-free and overall survival
      * If they failed to achieve CR/CRi, they are assessable for response, event-free, and overall survival
2. Performance status ≤ 3 (Eastern Cooperative Oncology Group [ECOG] Scale)
3. Adequate liver and renal function as defined by the following criteria:

   * Total serum bilirubin ≤ 1.5 x upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) ≤ 3 x ULN, unless due to disease involvement of the liver or hemolysis, in which case an ALT ≤ 10 x ULN is acceptable
   * Aspartate aminotransferase (AST) ≤ 3 x ULN, unless due to disease involvement of the liver or hemolysis, in which case an ALT ≤ 10 x ULN is acceptable
   * Creatinine clearance ≥ 30 mL/min
   * INR ≤ 1.5 x ULN and aPTT . 1.5 x ULN
4. For females of childbearing potential, a negative pregnancy test must be documented within 1 week of starting treatment
5. Female and male patients who are fertile must agree to use an effective form of contraception (birth control methods while on study, such as birth control pills or injections, intrauterine devices [IUDs]), or double-barrier methods (for example, a condom in combination with spermicide) with their sexual partners for 4 months after the end of treatment
6. Signed informed consent

Exclusion Criteria:

1. Patients with Philadelphia chromosome-positive ALL or Burkitt leukemia
2. Patients who are willing and eligible to receive intensive chemotherapy (only for patients enrolling in frontline cohort)
3. Active serious infection not controlled by oral or intravenous antibiotics
4. Known CNS leukemia requiring radiation
5. Active GVHD
6. Active secondary malignancy other than skin cancer (e.g., basal cell carcinoma or squamous cell carcinoma) that in the investigator's opinion will shorten survival to less than 1 year
7. Known hepatitis B or C infection, or known seropositivity for human immunodeficiency virus (HIV)
8. Active grade III-V cardiac failure as defined by the New York Heart Association Criteria
9. Patients with a cardiac ejection fraction (as measured by either multigated acquisition [MUGA] or echocardiogram) < 40%
10. Received moderate or strong CYP3A inhibitors or strong CYP3A inducers within 7 days of starting venetoclax
11. Received medication that interferes with coagulation or platelet function within 7 days prior to the first dose of study drug or during the study treatment period
12. Consumed grapefruit, grapefruit products, Seville oranges, or star fruit within 3 days prior to starting venetoclax
13. Prior history of treatment with navitoclax.
14. Treatment with any investigational antileukemic agents or chemotherapy agents in the last 7 days before study entry, unless full recovery from side effects has occurred or patient has rapidly progressive disease judged to be life-threatening by the investigator. Exception: Treatment with hydroxyurea and/or dexamethasone are allowed prior to study treatment, without window of exclusion
15. Pregnant and lactating women will not be eligible; women of childbearing potential should have a negative pregnancy test prior to entering on the study and be willing to practice methods of contraception. Women do not have childbearing potential if they have had a hysterectomy or are postmenopausal without menses for 12 months. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control
16. History of significant bleeding disorder unrelated to cancer, including: diagnosed congenital bleeding disorders (e.g., von Willebrand's disease); diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
17. Patient with total serum bilirubin > 1.5 x upper limit of normal (ULN).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-04-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (Phase I) | Up to 28 days
  The MTD is the highest dose level in which < 2 patients of 6 develop first cycle dose-limiting toxicity (DLT).
DLT (Phase I) | Up to 28 days
  A non-hematologic DLT is defined as a clinically significant (as assessed by treating physician) grade 3 or 4 adverse event or abnormal laboratory value (according to Common Terminology Criteria for Adverse Events [CTCAE] criteria). Toxicity type, severity and attribution will be summarized for each patient using frequency tables.

SECONDARY OUTCOMES:
Overall response rate (Phase II) | Up to 56 days (2 courses)
  Will be defined as the percentage of patients achieving a complete response (CR) or CR with inadequate count recovery (CRi). Will estimate the overall response (OR) for the combination treatment, along with the 95% credible interval.
Minimal residual disease (MRD) negativity | Up to 4 years
  Will be summarized using descriptive statistics such as mean, standard deviation, median and range.
Duration of response (DOR) | Up to 4 years
  Will be summarized using descriptive statistics such as mean, standard deviation, median and range. The association between response and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Event-free survival (EFS) | From the first day of treatment until any failure (resistant disease, relapse, or death), assessed up to 4 years
  The association between response and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Overall survival (OS) | From the first day of treatment to time of death from any cause, assessed up to 4 years
  The association between response and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Incidence of adverse events | Up to 4 years
  Will be summarized using descriptive statistics such as mean, standard deviation, median and range.

OTHER OUTCOMES:
Apoptotic protein expression and Bcl-2 dependency | Up to 4 years
  Apoptotic protein expression and Bcl-2 dependency will be correlated on response and resistance to the combination regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Elias Jabbour, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Short NJ, Jabbour E, Jain N, Senapati J, Nasr L, Haddad FG, Li Z, Hsiao YC, Yang JJ, Pemmaraju N, Ohanian M, Wierda WG, Montalban-Bravo G, Borthakur G, Han L, Xiao L, Huang X, Abramova R, Zhao M, Garris R, Konopleva M, Ravandi F, Kantarjian H. A phase 1/2 study of mini-hyper-CVD plus venetoclax in patients with relapsed/refractory acute lymphoblastic leukemia. Blood Adv. 2024 Feb 27;8(4):909-915. doi: 10.1182/bloodadvances.2023012231. PMID 38207208
- See also: MD Anderson Cancer Center — http://www.mdanderson.org